CLINICAL TRIAL: NCT02840279
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Examine the Safety, Tolerability, Pharmacokinetic, and Preliminary Cognitive Profile of BPN14770 in Healthy Young and Elderly Male and Female Subjects
Brief Title: A Multiple Ascending Dose Study of BPN14770 in Healthy Young and Elderly Male or Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPN14770-CNS-102
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: cognition; dementia; phosphodiesterase type 4D; PDE4D
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPN14770 (Experimental): An oral dose of BPN14770
  Interventions: Drug: BPN14770
- Placebo (Placebo Comparator): An oral dose of placebo matching BPN14770
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPN14770 — BPN14770 is an investigational new drug being developed for the treatment of Alzheimer's disease and other cognitive disorders. BPN14770 is a small molecule, subtype selective, negative allosteric modulator of phosphodiesterase 4D.
  Arms: BPN14770
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind (Investigator and subject-blinded) placebo-controlled, multiple, ascending-dose study to evaluate the safety, tolerability, and pharmacokinetic profile of BPN14770 in healthy young and elderly male and female subjects and to provide a preliminary assessment of the cognitive effects of BPN14770 in healthy elderly subjects.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the safety and tolerability profile of multiple oral ascending dose levels of BPN14770 in healthy young and elderly subjects.
2. To characterize the plasma pharmacokinetic profile of BPN14770 following oral administration in healthy young and elderly subjects.
3. To provide preliminary assessment of the cognitive effect of BPN14770 in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy young males or females between the ages of 21 to 45, inclusive (Cohorts 1, 2, 3 and 7; female subjects must not be pregnant or breastfeeding), and healthy elderly males or females ≥ 65 years of age (Cohorts 4, 5, 6).
2. Body mass index between 18 kg/m2 to 32 kg/m2, inclusive, and body weight of ≥50 kg (110 pounds).
3. Female subjects must be surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to dosing), at least two years post-menopausal, or willing to use two barrier methods of contraception from initial screening until one month after taking the last dose of study drug. Barrier methods of contraception include diaphragm, cervical cap, male condom, female condom, and spermicidal foam and sponges. Menopausal status declared by females in the young cohorts will be verified by a follicle stimulating hormone (FSH) test at Screening. In addition, all females must have a negative pregnancy test within 48 hours before dosing on Day 1 regardless of childbearing potential.
4. Male subjects must be willing to inform female partners of their participation in the study and must agree to use adequate contraceptive methods (vasectomy performed at least 6 months prior to dosing or use at least one barrier method of birth control).
5. Able to understand the study procedures, voluntarily consent to participate in this study, and provide written informed consent prior to start of any study-specific procedures.
6. Willing and able to remain in the study unit for the entire duration of the confinement period, and return for outpatient visits.

Exclusion Criteria:

1. Clinically significant abnormality, in the Investigator's judgement, indicated by the current hematology, biochemistry, or urinalysis tests, or from medical history, social history, vital signs, or physical examination.
2. Positive serology results for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
3. Marked hypotension (systolic blood pressure [BP] ˂90 mmHg or diastolic BP ˂50 mmHg) or hypertension (systolic BP ˃150 mmHg or diastolic BP ˃100 mmHg) based on supine and sitting values obtained at Screening, Day-1, or Day 1 predose. Out-of-range vital signs may be repeated once during each eligibility assessment (prior to the start of dosing on Day 1).
4. Marked bradycardia (heart rate ˂45 beats per minute [bpm]) or tachycardia (heart rate ˃110 bpm) based on supine ECG values obtained at Screening, Day -1, or Day 1 predose. Out-of-range vital signs may be repeated once at each eligibility assessment (prior to the start of dosing on Day 1).
5. Current or past history of significant (in the Investigator's judgement) cardiovascular, cerebrovascular, pulmonary, renal, or liver disease. Stable, well-controlled hypertension and hyperlipidemias are allowed (see Exclusion #10).
6. History of hematological disorders (e.g., thrombocytopenia) in the immediate family (i.e., parents and siblings).
7. Clinically important or significant conduction abnormalities on single ECG (including QTc interval ˃450 msec) or evidence or history of long QT syndrome. This exclusion applies to the ECGs obtained at Screening, Day -1, and Day 1 predose.
8. Current or past history of gastric or duodenal ulcers or other diseases of the gastrointestinal tract that could interfere with absorption of study drug. Note: Subjects with a history of appendectomy or cholecystectomy may be enrolled.
9. Active acute or chronic infectious diseases.
10. Unable to discontinue medications including psychotropic drugs, sedative antihistamines, or other centrally active medications [e.g., CNS beta blockers], and moderate to strong inhibitors or inducers of CYP3A4, CYP2D6, or other cytochromes). Other prescription or non-prescription drugs such as antihypertensive or cholesterol lowering drugs are allowed if, in the Investigator's judgement, they would not interfere with the test medication or the cognitive testing.
11. Any history of alcohol or drug abuse within the previous year prior to the Screening visit (per the current edition of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5), or regular (daily) consumption of alcohol exceeding two bottles of beer, or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
12. Any use of alcohol within 24 hours of admission into the study on Day -2.
13. Active smokers or tobacco users (e.g., chew and snuff) who are unable to discontinue tobacco use at least 3 months prior to admission to the study on Day -2 and refrain from using tobacco during the study treatment and evaluation period.
14. Inability or unwillingness to comply with the protocol, or likely inability to complete the study.
15. Participation in other clinical studies involving investigational drug within the previous 30 days prior to the Screening visit.
16. Donation of blood or blood products (including plasma) during the 8 weeks before the first administration of study drug on Day 1.
17. Positive screen for drugs of abuse or cotinine (at screen or upon admission), or a positive alcohol result (upon admission).
18. History of allergy to penicillin or sulfonamides, or any other clinically significant drug allergy that includes symptoms such as shortness of breath, rash, or edema.
19. Inability or unwillingness to perform the tasks necessary for the CogState Cognitive Function Assessments (elderly cohorts).
20. A suicidal ideation intensity score of 2 or higher per screening C-SSRS assessment and/or any suicidal behavior within the past 30 days.

Cognitive Testing Criteria:

Eligibility requirements for subjects in the elderly cohorts include successful completion of a computerized battery of CogState cognitive function assessments, including:

* Detection Task (DET)
* Identification Task (IDN)
* One Card Learning Task (OCL)
* One Back Task (ONB)
* Continuous Paired Associate Learning (CPAL)
* International Shopping List Task (ISLT)
* Groton Maze Learning Test (GMLT)

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 weeks
  Incidence and nature of adverse events (AEs) and serious adverse events (SAEs). Significant assessments reported as AEs or SAEs include clinical laboratory assessments and vital signs, physical and neurological examination, 12-lead electrocardiogram (ECG)

SECONDARY OUTCOMES:
Area Under the Curve from Time Zero to Twelve Hours [AUC0-12] | 2 weeks
Area Under the Concentration Time Curve from Zero to 12 Hours, Corrected for Dose [AUC12/D] | 2 weeks

OTHER OUTCOMES:
ISLT-D | 2 weeks
  International Shopping List Test words recalled at 24 hours
GMLT-D | 2 weeks
  Groton Maze Learning Test errors at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reines, MD, PhD, Study Chair — Tetra Discovery Partners
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowie JM, Gurney ME. The Use of Facebook Advertising to Recruit Healthy Elderly People for a Clinical Trial: Baseline Metrics. JMIR Res Protoc. 2018 Jan 24;7(1):e20. doi: 10.2196/resprot.7918. PMID 29367186